CLINICAL TRIAL: NCT02525679
Title: Single-blind, Partially Randomised, Placebo-controlled Phase I Study to Investigate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Rising Intravenous Doses of BI 655130 in Healthy Male Volunteers
Brief Title: Study to Investigate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of BI 655130 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1368.1; 2015-001931-19 (EudraCT Number)
Record Dates: First submitted 2015-08-14; First posted 2015-08-17 (Estimated); Results first posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2023-09

CONDITIONS: Healthy
MeSH Terms: interventions — spesolimab

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BI 655130 (spesolimab) (Experimental)
  Interventions: Drug: BI 655130 (spesolimab)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 655130 (spesolimab)
  Arms: BI 655130 (spesolimab)
Drug: Placebo
  Arms: Placebo

SUMMARY:
The aim of this study is to investigate the safety and tolerability of BI 655130 in healthy male subjects following single rising low, medium and high doses.

ELIGIBILITY:
Inclusion criteria:

* Healthy male subjects according to the investigators assessment, based on a complete medical history including a physical examination, vital signs (BP - Blood Pressure, PR - Puls Rate), 12-lead ECG (Electrocardiogram), and clinical laboratory tests
* Age of 18 to 45 years (incl.)
* BMI (Body Mass Index) of 18.5 to 29.9 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with GCP and local legislation

Exclusion criteria:

* Any finding in the medical examination (including BP - Blood Pressure, PR - Pulse Rate or ECG - Electrocardiogram) is deviating from normal and judged as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy and/or surgery of the gastrointestinal tract (except appendectomy and simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* Further exclusion criteria apply

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2015-09-14 (Actual); Primary Completion 2016-05-27 (Actual); Study Completion 2016-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- SGS Life Science Services - Clinical Research, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- [Derived] Joseph D, Thoma C, Haeufel T, Li X. Assessment of the Pharmacokinetics and Safety of Spesolimab, a Humanised Anti-interleukin-36 Receptor Monoclonal Antibody, in Healthy Non-Japanese and Japanese Subjects: Results from Phase I Clinical Studies. Clin Pharmacokinet. 2022 Dec;61(12):1771-1787. doi: 10.1007/s40262-022-01176-5. Epub 2022 Dec 1. PMID 36451029
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 78 subjects were randomised to 11 sequential dose groups (including an unplanned dose group). All subjects completed the trial according to the protocol. 3 subjects were not dosed as planned: they received 0.050 mg/kg BI 655130 instead of the planned 0.100 mg/kg BI 655130.
Pre-assignment Details: A total of 80 subjects were planned to be included in 10 sequential dose groups, each consisting of 8 subjects (6 on BI 655130 and 2 on placebo). However, 1 additional dose group was introduced to accommodate for a dosing error administration of 0.050 mg/kg instead of 0.100 mg/kg;
Groups:
- 0.001 mg/kg BI 655130 (Dose Group 1): Male healthy volunteers received single dose of 0.001 milligrams/kilograms (mg/kg) BI 655130 as concentrate for solution for Intravenous (IV) 30 min infusion
- 0.003 mg/kg BI 655130 (Dose Group 2): Male healthy volunteers received single dose of 0.003 mg/kg BI 655130 as concentrate for solution for IV 30 min infusion
- 0.010 mg/kg BI 655130 (Dose Group 3): Male healthy volunteers received single dose of 0.010 mg/kg BI 655130 as concentrate for solution for IV 30 min infusion
- 0.030 mg/kg BI 655130 (Dose Group 4): Male healthy volunteers received single dose of 0.030 mg/kg BI 655130 as concentrate for solution for IV 30 min infusion
- 0.100 mg/kg BI 655130 (Dose Group 5): Male healthy volunteers received single dose of 0.100 mg/kg BI 655130 as concentrate for solution for IV 30 min infusion
- 0.300 mg/kg BI 655130 (Dose Group 6): Male healthy volunteers received single dose of0.300 mg/kg BI 655130 as concentrate for solution for IV 30 min infusion
- 1 mg/kg BI 655130 (Dose Group 7): Male healthy volunteers received single dose of 1 mg/kg BI 655130 as concentrate for solution for IV 30 min infusion
- 3 mg/kg BI 655130 (Dose Group 8): Male healthy volunteers received single dose of 3 mg/kg BI 655130 as concentrate for solution for IV 30 min infusion
- 6 mg/kg BI 655130 (Dose Group 9): Male healthy volunteers received single dose of 6 mg/kg BI 655130 as concentrate for solution for IV 30 min infusion
- 10 mg/kg BI 655130 (Dose Group 10): Male healthy volunteers received single dose of 10 mg/kg BI 655130 as concentrate for solution for IV 30 min infusion
- 0.050 mg/kg BI 655130 (Unplanned): Male healthy volunteers received single dose of 0.050 mg/kg BI 655130 as concentrate for solution for IV 30 min infusion (unit strength: 20 milligrams/milliLitres (mg/mL). This separate group (unplanned) was introduced to accommodate subjects who had been wrongly administered 0.050 mg/kg BI 655130 instead of the planned 0.100 mg/kg BI 655130
- Placebo: Male healthy volunteers received single dose of matching placebo as concentrate for solution for IV 30 min infusion.
Period: Overall Study
Arm/Group | 0.001 mg/kg BI 655130 (Dose Group 1) | 0.003 mg/kg BI 655130 (Dose Group 2) | 0.010 mg/kg BI 655130 (Dose Group 3) | 0.030 mg/kg BI 655130 (Dose Group 4) | 0.100 mg/kg BI 655130 (Dose Group 5) | 0.300 mg/kg BI 655130 (Dose Group 6) | 1 mg/kg BI 655130 (Dose Group 7) | 3 mg/kg BI 655130 (Dose Group 8) | 6 mg/kg BI 655130 (Dose Group 9) | 10 mg/kg BI 655130 (Dose Group 10) | 0.050 mg/kg BI 655130 (Unplanned) | Placebo
Started | 6 | 6 | 6 | 6 | 5 | 4 | 6 | 6 | 6 | 4 | 3 | 20
Completed | 6 | 6 | 6 | 6 | 5 | 4 | 6 | 6 | 6 | 4 | 3 | 20
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The TS included all subjects from the randomised set who were documented to have taken at least 1 dose of trial medication. All 78 randomised subjects were included in the TS.
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.001 mg/kg BI 655130 (Dose Group 1) | 0.003 mg/kg BI 655130 (Dose Group 2) | 0.010 mg/kg BI 655130 (Dose Group 3) | 0.030 mg/kg BI 655130 (Dose Group 4) | 0.100 mg/kg BI 655130 (Dose Group 5) | 0.300 mg/kg BI 655130 (Dose Group 6) | 1 mg/kg BI 655130 (Dose Group 7) | 3 mg/kg BI 655130 (Dose Group 8) | 6 mg/kg BI 655130 (Dose Group 9) | 10 mg/kg BI 655130 (Dose Group 10) | 0.050 mg/kg BI 655130 (Unplanned) | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 4 | 6 | 6 | 6 | 4 | 3 | 20 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.5 (5.0) | 33.2 (8.1) | 33.2 (8.7) | 31.2 (8.0) | 40.0 (2.5) | 33.5 (2.6) | 32.5 (7.7) | 34.2 (6.5) | 36.0 (9.9) | 29.8 (5.6) | 31.0 (7.0) | 34.2 (8.5) | 33.1 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 6 | 6 | 6 | 6 | 5 | 4 | 6 | 6 | 6 | 4 | 3 | 20 | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 6 | 6 | 6 | 6 | 4 | 4 | 6 | 6 | 6 | 4 | 3 | 20 | 77
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 6 | 6 | 6 | 6 | 5 | 4 | 6 | 5 | 6 | 4 | 3 | 19 | 76
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 00 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Drug Related Adverse Events
Description: Percentage of subjects with drug related adverse events are presented.
Time Frame: Adverse events reported until the end-of-trial examination; up to day 74
Population: Treated set
Measure: Number; unit: percentage of participants
Arm/Group | 0.001 mg/kg BI 655130 (Dose Group 1) | 0.003 mg/kg BI 655130 (Dose Group 2) | 0.010 mg/kg BI 655130 (Dose Group 3) | 0.030 mg/kg BI 655130 (Dose Group 4) | 0.100 mg/kg BI 655130 (Dose Group 5) | 0.300 mg/kg BI 655130 (Dose Group 6) | 1 mg/kg BI 655130 (Dose Group 7) | 3 mg/kg BI 655130 (Dose Group 8) | 6 mg/kg BI 655130 (Dose Group 9) | 10 mg/kg BI 655130 (Dose Group 10) | 0.050 mg/kg BI 655130 (Unplanned) | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 4 | 6 | 6 | 6 | 4 | 3 | 20
percentage of participants | 16.7 | 16.7 | 33.3 | 0.0 | 0.0 | 0.0 | 16.7 | 0.0 | 33.3 | 0.0 | 33.3 | 15.0

2. Secondary Outcome: Maximum Measured Concentration of BI 655130 in Plasma (Cmax)
Description: Maximum measured concentration of BI 655130 in plasma (Cmax) is presented.
Time Frame: -2 hours (h) before and 0.5h, 1h, 2h, 3h, 4h, 8h, 12h, 24h, 48h, 72h, 96h, 168h, 336h, 504h, 672h, 840h, 1008h, 1344h, 1680h after drug administration
Population: Descriptive pharmacokinetic analysis set (PKSD): The descriptive analysis of PK (pharmacokinetic) concentrations and parameters was based on all treated subjects who provided at least 1 PK concentration (plasma or urine) that was judged as PK evaluable and not affected by protocol violations relevant to the evaluation of PK parameters.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/milliLitres (μg/mL)
Arm/Group | 0.001 mg/kg BI 655130 (Dose Group 1) | 0.003 mg/kg BI 655130 (Dose Group 2) | 0.010 mg/kg BI 655130 (Dose Group 3) | 0.030 mg/kg BI 655130 (Dose Group 4) | 0.100 mg/kg BI 655130 (Dose Group 5) | 0.300 mg/kg BI 655130 (Dose Group 6) | 1 mg/kg BI 655130 (Dose Group 7) | 3 mg/kg BI 655130 (Dose Group 8) | 6 mg/kg BI 655130 (Dose Group 9) | 10 mg/kg BI 655130 (Dose Group 10) | 0.050 mg/kg BI 655130 (Unplanned)
Number analyzed (Participants) | 6 | 6 | 4 | 6 | 5 | 4 | 6 | 6 | 6 | 4 | 3
micrograms/milliLitres (μg/mL) | NA (NA) — Not available as plasma concentrations were below lower limit of quantification (BLQ) | NA (NA) — Not available as plasma concentrations were below lower limit of quantification (BLQ) | 0.0228 (33.5) | 0.413 (21.2) | 1.96 (11.9) | 6.63 (3.28) | 20.3 (13.6) | 60.6 (7.17) | 153 (12.7) | 235 (2.79) | 0.998 (15.7)
Statistical Analysis 1: Comparison: 0.010 mg/kg BI 655130 (Dose Group 3) vs 0.030 mg/kg BI 655130 (Dose Group 4) vs 0.100 mg/kg BI 655130 (Dose Group 5) vs 0.300 mg/kg BI 655130 (Dose Group 6); Dose proportionality in plasma for Cmax (log-transformed scale) was explored based on the linear regression model; Test type: Superiority or Other; Slope = 1.5968, 95% CI 2-sided [1.3784 to 1.8151], Standard Error of Mean 0.1047 — Based on the estimate for the slope parameter, a two sided 95% confidence interval for the slope was computed. Perfect dose proportionality would correspond to a slope of 1. Standard error (SE) of the mean is actually SE of the slope
Statistical Analysis 2: Comparison: 0.300 mg/kg BI 655130 (Dose Group 6) vs 1 mg/kg BI 655130 (Dose Group 7) vs 3 mg/kg BI 655130 (Dose Group 8) vs 6 mg/kg BI 655130 (Dose Group 9) vs 10 mg/kg BI 655130 (Dose Group 10); Dose proportionality in plasma for Cmax (log-transformed scale) was explored based on the linear regression model; Test type: Superiority or Other; Slope = 1.0207, 95% CI 2-sided [0.9668 to 1.0747], Standard Error of Mean 0.0261 — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Area Under the Concentration-time Curve of the BI 655130 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of the BI 655130 in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) is presented.
  Reliable values of AUC0-∞ could not be calculated because concentrations were too high at the last PK sample collected "1680h" after drug administration. AUC0-tz was utilized for the dose proportionality analyses instead of AUC0-∞.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms*day/milliLitres (μg*day/mL)
Arm/Group | 0.001 mg/kg BI 655130 (Dose Group 1) | 0.003 mg/kg BI 655130 (Dose Group 2) | 0.010 mg/kg BI 655130 (Dose Group 3) | 0.030 mg/kg BI 655130 (Dose Group 4) | 0.100 mg/kg BI 655130 (Dose Group 5) | 0.300 mg/kg BI 655130 (Dose Group 6) | 1 mg/kg BI 655130 (Dose Group 7) | 3 mg/kg BI 655130 (Dose Group 8) | 6 mg/kg BI 655130 (Dose Group 9) | 10 mg/kg BI 655130 (Dose Group 10) | 0.050 mg/kg BI 655130 (Unplanned)
Number analyzed (Participants) | 6 | 6 | 4 | 6 | 5 | 4 | 6 | 6 | 6 | 4 | 3
micrograms*day/milliLitres (μg*day/mL) | NA (NA) — Not available as plasma concentrations were below lower limit of quantification (BLQ) | NA (NA) — Not available as plasma concentrations were below lower limit of quantification (BLQ) | 0.0234 (125) | 2.35 (23.9) | 27.7 (16.6) | 127 (6.05) | 563 (26.2) | 1260 (6.81) | 3380 (15.6) | 5080 (18.9) | 13.0 (6.59)

4. Secondary Outcome: Area Under the Concentration-time Curve of the BI 655130 in Plasma Over the Time Interval From 0 to the Last Measurable Plasma Concentration (AUC0-tz)
Description: Area under the concentration-time curve of the BI 655130 in plasma over the time interval from 0 to the last measurable plasma concentration (AUC0-tz) is presented.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms*day/milliLitres (μg*day/mL)
Arm/Group | 0.001 mg/kg BI 655130 (Dose Group 1) | 0.003 mg/kg BI 655130 (Dose Group 2) | 0.010 mg/kg BI 655130 (Dose Group 3) | 0.030 mg/kg BI 655130 (Dose Group 4) | 0.100 mg/kg BI 655130 (Dose Group 5) | 0.300 mg/kg BI 655130 (Dose Group 6) | 1 mg/kg BI 655130 (Dose Group 7) | 3 mg/kg BI 655130 (Dose Group 8) | 6 mg/kg BI 655130 (Dose Group 9) | 10 mg/kg BI 655130 (Dose Group 10) | 0.050 mg/kg BI 655130 (Unplanned)
Number analyzed (Participants) | 6 | 6 | 4 | 6 | 5 | 4 | 6 | 6 | 6 | 4 | 3
micrograms*day/milliLitres (μg*day/mL) | NA (NA) — Not available as plasma concentrations were below lower limit of quantification (BLQ) | NA (NA) — Not available as plasma concentrations were below lower limit of quantification (BLQ) | 0.00652 (121) | 2.08 (29.0) | 25.1 (15.5) | 113 (5.86) | 420 (13.3) | 1050 (7.26) | 2610 (11.7) | 4130 (12.1) | 9.57 (5.90)
Statistical Analysis 1: Comparison: 0.010 mg/kg BI 655130 (Dose Group 3) vs 0.030 mg/kg BI 655130 (Dose Group 4) vs 0.100 mg/kg BI 655130 (Dose Group 5) vs 0.300 mg/kg BI 655130 (Dose Group 6); Dose proportionality in plasma for AUC(0-tz) (log-transformed scale) was explored based on the linear regression model; Test type: Superiority or Other; Slope = 2.7123, 95% CI 2-sided [2.1856 to 3.2389], Standard Error of Mean 0.2525 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: 0.300 mg/kg BI 655130 (Dose Group 6) vs 1 mg/kg BI 655130 (Dose Group 7) vs 3 mg/kg BI 655130 (Dose Group 8) vs 6 mg/kg BI 655130 (Dose Group 9) vs 10 mg/kg BI 655130 (Dose Group 10); Dose proportionality in plasma for AUC(0-tz) (log-transformed scale) was explored based on the linear regression model; Test type: Superiority or Other; Slope = 1.0003, 95% CI 2-sided [0.9482 to 1.0525], Standard Error of Mean 0.0253 — [estimate comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse events reported until the end-of-trial examination; up to day 74.
Description: Treated set (TS): The TS included all subjects from the randomised set who were documented to have taken at least 1 dose of trial medication. All 78 randomised subjects were included in the TS.
Arm/Group | Placebo | 0.001 mg/kg BI 655130 (Dose Group 1) | 0.003 mg/kg BI 655130 (Dose Group 2) | 0.010 mg/kg BI 655130 (Dose Group 3) | 0.030 mg/kg BI 655130 (Dose Group 4) | 0.100 mg/kg BI 655130 (Dose Group 5) | 0.300 mg/kg BI 655130 (Dose Group 6) | 1 mg/kg BI 655130 (Dose Group 7) | 3 mg/kg BI 655130 (Dose Group 8) | 6 mg/kg BI 655130 (Dose Group 9) | 10 mg/kg BI 655130 (Dose Group 10) | 0.050 mg/kg BI 655130 (Unplanned)
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/6 | 0/6 | 0/6 | 0/6 | 0/5 | 0/4 | 0/6 | 0/6 | 0/6 | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 11/20 | 2/6 | 4/6 | 5/6 | 5/6 | 4/5 | 2/4 | 5/6 | 3/6 | 3/6 | 1/4 | 2/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=20) | 0.001 mg/kg BI 655130 (Dose Group 1) (N=6) | 0.003 mg/kg BI 655130 (Dose Group 2) (N=6) | 0.010 mg/kg BI 655130 (Dose Group 3) (N=6) | 0.030 mg/kg BI 655130 (Dose Group 4) (N=6) | 0.100 mg/kg BI 655130 (Dose Group 5) (N=5) | 0.300 mg/kg BI 655130 (Dose Group 6) (N=4) | 1 mg/kg BI 655130 (Dose Group 7) (N=6) | 3 mg/kg BI 655130 (Dose Group 8) (N=6) | 6 mg/kg BI 655130 (Dose Group 9) (N=6) | 10 mg/kg BI 655130 (Dose Group 10) (N=4) | 0.050 mg/kg BI 655130 (Unplanned) (N=3)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 2 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Injection site haematoma (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 3 | 0 | 0 | 1 | 4 | 2 | 0 | 1 | 2 | 1 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 3 | 1 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.